CLINICAL TRIAL: NCT03067571
Title: An Open-Label, Phase 2 Trial Evaluating the Efficacy and Safety of Daratumumab in Subjects With Relapsed/Refractory Acute Myelogenous Leukemia or High-Risk Myelodysplastic Syndrome
Brief Title: Daratumumab in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated early because of lack of efficacy
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0889; NCI-2018-01222 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0889 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-02-24; First posted 2017-03-01 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: High Risk Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (daratumumab) (Experimental): Patients receive daratumumab IV over 3.25-6.5 hours on days 1, 8, 15 and 22 of cycles 1-2, on days 1 and 15 of cycles 3-6, and on day 1 of subsequent cycles. Cycles repeat every 28 days.
  Interventions: Biological: Daratumumab

INTERVENTIONS:
Biological: Daratumumab — Given IV
  Other Names: Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414

SUMMARY:
This phase II trial studies how well daratumumab works in treating patients with acute myeloid leukemia that has come back or does not respond to treatment or high-risk myelodysplastic syndrome. Immunotherapy with monoclonal antibodies, such as daratumumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
The goal of this clinical research study is to learn if daratumumab in combination with venetoclax can help to control acute myelogenous leukemia (AML), high-risk myelodysplastic syndrome (MDS) that is refractory (does not respond to treatment) or relapsed (comes back after being treated), or relapsed/refractory T acute lymphoblastic leukemia/lymphoma (T-ALL, T-LBL) .

OUTLINE:

Patients receive daratumumab intravenously (IV) over 3.25-6.5 hours on days 1, 8, 15 and 22 of cycles 1-2, on days 1 and 15 of cycles 3-6, and on day 1 of subsequent cycles. Cycles repeat every 28 days.

After completion of study treatment, patients are followed up monthly for 1 year, every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Age >/=18 years at the time of signing the informed consent form
* Diagnosis of AML [other than acute promyelocytic leukemia (APL)] with refractory/relapsed disease; patients with relapsed/refractory high-risk [(intermediate-2 or higher by International Prognostic Scoring System (IPSS) and/or >/= 10% blasts)] MDS will also be eligible. (Treatment approach for relapsed/refractory AML is very similar to that of high risk MDS), or diagnosis of relapsed/refractory T-ALL/T-LBL.
* All non-hematological toxicity of previous cancer therapy should have resolved to =< grade 1 (except alopecia or other toxicities not involving major organs)
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2 at study entry
* Serum creatinine </= 2 mg/dL and estimated glomerular filtration rate or creatinine clearance >/= 40 ml/min
* Total bilirubin =< 2 mg/dL
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) =< 3 x upper limit of normal (ULN)
* Women of childbearing potential must be practicing a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies: eg, established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device or intrauterine system; barrier methods: condom with spermicidal foam/gel/film/cream/suppository or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository; male partner sterilization (the vasectomized partner should be the sole partner for that subject); true abstinence (when this is in line with the preferred and usual lifestyle of the subject) during and after the study (3 months after the last dose of daratumumab for women)
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control eg, either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 3 months after receiving the last dose of study drug
* AML relapse > 6 months since autologous or allogeneic stem cell transplantation, provided there is no active graft-versus-host disease (GVHD) > grade 1; no treatment with high dose steroids for GVHD (up to 20 mg prednisolone or equivalent); no treatment with immunosuppressive drugs with the exception of low dose cyclosporine and tacrolimus (blood levels of 0.5-0.6 ug/mL)

Exclusion Criteria:

* White blood cell count more than 25 × 109 /L prior to initiation of venetoclax
* Pregnant or breast feeding females
* Cancer chemotherapy within 2 weeks prior to start of daratumumab treatment (exception hydroxyurea). Use of hydroxyurea to control proliferative disease will be allowed prior to starting therapy on study and for 7 days during cycle 1-3 (maximum daily dose of 7 gm)
* Subject has received daratumumab or other anti-CD38 therapies previously
* Subject has received a cumulative dose of corticosteroids more than the equivalent of >= 140 mg of prednisone within the 2 week period before cycle 1, day 1
* Subject has known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal. NOTE: FEV1 testing is required for patients suspected of having COPD and subjects must be excluded if FEV1 < 50% of predicted normal
* Subject has a history of another malignancy within 5 years before cycle 1, day 1 (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the investigator, with concurrence with the IND office and supporter's medical monitor, is considered cured with minimal risk of recurrence)
* Subject is known to be seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti- HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR
* Subjects who are seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy) will be excluded.
* Subject has clinically significant cardiac disease, including: myocardial infarction within 1 year before Cycle 1, Day 1, or unstable or uncontrolled disease/condition related to or affecting cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV); cardiac arrhythmia (Common Terminology Criteria for Adverse Events [CTCAE] version 4.03 grade 2 or higher) or clinically significant electrocardiogram (ECG) abnormalities; screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) > 470 msec
* Subject has known severe allergies, hypersensitivity, or intolerance to monoclonal antibodies or human proteins, or their excipients (refer to the latest version of the Investigator Brochure), or known sensitivity to mammalian-derived products
* Subject has any concurrent medical condition or disease (eg, active systemic infection, laboratory abnormalities) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study
* Exclude patients with known Kell antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Daratumumab)
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Daratumumab)
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 68 [38 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Participants With a Response
Description: Response rate as determined by the International Working Group recommendations. Complete remission (CR): The patient must be free of all symptoms related to leukemia and have an absolute neutrophil count >/= 1.0 x 109/L, platelet count >/- 100 x 109/L, and normal bone marrow differential (</= 5% blasts). Complete remission without platelet recovery (CRp): As per CR but platelet count < 100 x 109/L. Partial remission (PR): CR with 6 to 25% abnormal cells in the marrow or 50% decrease in bone marrow blasts. Marrow CR: Bone marrow: </= 5% myeloblasts and decrease by >/= 50% over pre-treatment (MDS only). Morphologic leukemia-free state: Normal marrow differential (<5% blasts); absolute neutrophil count and platelet counts are not considered. (AML only). Hematologic Improvement (HI): HI should be described by the number of individual, positively affected cell lines
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Daratumumab): Patients receive daratumumab IV over 3.25-6.5 hours on days 1, 8, 15 and 22 of cycles 1-2, on days 1 and 15 of cycles 3-6, and on day 1 of subsequent cycles. Cycles repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Daratumumab: Given IV
Arm/Group | Treatment (Daratumumab)
Number analyzed (Participants) | 7
Participants | 0

2. Secondary Outcome: Time on Treatment
Description: Time from date of start of study medication until date of off study.
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Daratumumab)
Number analyzed (Participants) | 7
Months | 1.1 [0.2 to 3.0]

3. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Daratumumab)
Number analyzed (Participants) | 7
Months | 4.2 [0.2 to 9.2]

4. Secondary Outcome: Progression Free Survival
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Daratumumab)
Number analyzed (Participants) | 7
Months | 1.1 [0.2 to 3.0]

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Treatment (Daratumumab)
All-Cause Mortality (participants affected / at risk) | 2/7
Serious Adverse Events (participants affected / at risk) | 6/7
Other Adverse Events (participants affected / at risk) | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Daratumumab) (N=7)
Angioedema (Immune system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile Neutropenia (Investigations) | 2 (2)
Infection (Infections and infestations) | 1 (1)
Lung Infection (Infections and infestations) | 1 (2)
Oral Mucositis (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Septic Shock (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Daratumumab) (N=7)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Fatigue (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/71/NCT03067571/Prot_SAP_000.pdf